CLINICAL TRIAL: NCT04817267
Title: Pilot Study of reSET-O to Treatment-as-usual in Acute Care Settings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ReSET-O product no longer available, Pear Therapeutics, Inc. filed for bankruptsy
Sponsor: Johns Hopkins University (Other)
Collaborators: Pear Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00282938
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reSET-O + Treatment-As-Usual (TAU) (Experimental): Participants randomly assigned to this group will receive the TAU plus the reSET-O app.
  Interventions: Device: reSET-O app
- Treatment-As-Usual (TAU) (No Intervention): Participants randomly assigned to this group will receive the TAU only (no use of the reSET-O app).

INTERVENTIONS:
Device: reSET-O app — The reSET-O app, a prescription digital therapeutic, provides cognitive behavioral therapy for opioid use disorder. The app provides psychoeducation related to opioid use, coping skills, and skills to avoid relapse.
  Arms: reSET-O + Treatment-As-Usual (TAU)

SUMMARY:
This randomized controlled pilot study will evaluate feasibility, acceptability, and potential efficacy of an app, reSET-O, for patients being started on buprenorphine in acute care settings.

DETAILED DESCRIPTION:
This randomized controlled pilot study will enroll 60 participants, who will be randomly assigned to a treatment as usual (TAU) group or a reSET-O+TAU group after being started on buprenorphine in acute care settings (e.g., emergency department) and referred to community treatment. Study enrollment will last for 3 months after discharge from the acute care setting. Participants in the reSET-O+TAU group will be provided with the reSET-O app and will be encouraged to engage with the app for the 3 months following discharge from the acute care unit. The app works as an extension of cognitive behavioral therapy, providing psychoeducation related to opioid use disorder. All participants will be assessed at study intake and every month during the 3-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Opioid use disorder
* Eligible for buprenorphine treatment
* Has reSET-O compatible mobile device

Exclusion Criteria:

* Pregnancy
* Significant psychiatric comorbidity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of approached patients who are eligible for and interested in participation | 3 months
  Percentage of approached patients who are eligible for and interested in participation will be used to assess feasibility.
Acceptability as assessed by the Treatment Acceptability Questionnaire | 3 months
  Participant responses to the Treatment Acceptability Questionnaire.
Acceptability as assessed by the System Usability Scale | 3 months
  Participant responses to the System Usability Scale.

SECONDARY OUTCOMES:
Attendance at follow-up appointment for on-going buprenorphine treatment within 30 days of discharge | 30 days
  Attendance at follow-up appointment for on-going buprenorphine treatment within 30 days of discharge will be used to assess Treatment Engagement.
Percentage of drug-negative urine samples during the 3-month intervention | 3 months
  Percentage of drug-negative urine samples during the 3-month intervention will be used to assess Illicit opioid/other drug use.

CONTACTS AND LOCATIONS:
Overall Officials: August Holtyn, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayivew Emergency Department, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No